CLINICAL TRIAL: NCT04544228
Title: Comparison of Effectiveness of Adding Ketamine or Neostigmine to Bupivacaine for Ultrasound Guided Serratus Anterior Plane Block in Modified Radical Mastectomy , Randomized Double Blinded Comparative Study.
Brief Title: Ketamine or Neostigmine for Serratus Anterior Plane Block in Modified Radical Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Bassant M. Abdelhamid, associate professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MS-101-2020
Record Dates: First submitted 2020-08-28; First posted 2020-09-10 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, General; Ketamine; Bupivacaine; Neostigmine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ketamine (Experimental): Patients will receive Ultrasound guided Serratus Anterior Plane Block preoperative with injection of 30 ml bupivacaine 0.25% + 1 ml ketamine
  Interventions: Procedure: Serratus Anterior Plane Block Technique; Procedure: General anesthesia; Drug: bupivacaine +ketamine
- Neostigmine (Experimental): Patients will receive Ultrasound guided Serratus Anterior Plane Block preoperative with injection of 30 ml bupivacaine 0.25% + 1 ml neostigmine
  Interventions: Procedure: Serratus Anterior Plane Block Technique; Procedure: General anesthesia; Drug: bupivacaine + neostigmine
- Control (Active Comparator): Patients will receive Ultrasound guided Serratus Anterior Plane Block preoperative with injection of 30 ml bupivacaine 0.25% + 1 ml normal saline.
  Interventions: Procedure: Serratus Anterior Plane Block Technique; Procedure: General anesthesia; Drug: bupivacaine +saline

INTERVENTIONS:
Procedure: Serratus Anterior Plane Block Technique — The patient will be placed in Lateral Decubitus with a surgical side upwards with arm abduction. A linear ultrasound transducer (6-13 MHz) will be placed on the patient's midaxillary line in the transverse plane, at the level of the fifth rib, with the indicator oriented toward the operator's left. With the rib, pleural line, and overlying serratus anterior and latissimus dorsi muscles visualized, local infiltration of the skin and subcutaneous tissue will be applied by 2-3ml of lidocaine 2%. Then, using ultrasound guidance, A 38-mm 22-gauge regional block needle will be advanced in-plane at an angle of approximately 45 degrees towards the fifth rib. The expecting depth for this block is 1-4 cm. After aspiration, injection 30ml local anesthetic mixture will be injected anteriorly to the rib and deep to the serratus anterior muscle.
Procedure: General anesthesia — Induction of general anaesthesia will be performed using a regimen of IV 2 μg/kg fentanyl and propofol IV 2 mg /kg. Tracheal intubation will be facilitated using 0.5 mg/kg IV of rocuronium.
  Anaesthesia will be maintained with inhaled sevoflurane 2-2.5% in oxygen enriched air (FiO2=0.5). Maintenance doses of rocuronium 0.1 m\kg will be provided every 30 minutes.
  The residual neuromuscular blockade will be reversed using neostigmine (0.05 mg/kg) and atropine (0.02 mg/kg), and extubation will be performed after complete recovery of the airway reflexes.
Drug: bupivacaine +ketamine — 30 ml bupivacaine 0.25% + 1 ml ketamine (50mg) in Serratus Anterior Plane Block.
  Other Names: ketamine
  Arms: ketamine
Drug: bupivacaine + neostigmine — 30 ml bupivacaine 0.25% + 1 ml neostigmine (500 μg)in Serratus Anterior Plane Block.
  Other Names: neostigmine
  Arms: Neostigmine
Drug: bupivacaine +saline — 30 ml bupivacaine 0.25% + 1 ml normal saline in Serratus Anterior Plane Block.
  Other Names: saline
  Arms: Control

SUMMARY:
The aim of this study is to Investigate the analgesic efficacy of adding ketamine compared to neostigmine to local anesthetic in Ultrasound guided Serratus anterior plane block for patients undergoing Modified Radical Mastectomy.

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy among females with incidence of 18,660 patients each year in Egypt. Modified Radical Mastectomy is considered the main surgical management for breast cancer accounting for 31% of all breast surgery cases.

Ultrasound guided Serratus anterior plane block provides analgesia for breast and lateral thoracic wall surgeries by blocking nerves that are located in a compartment between the serratus anterior and the latissimus dorsi muscles ( the intercostobrachial nerve, lateral cutaneous branches of the intercostal nerves (T3-T9), long thoracic nerve and thoracodorsal nerve).

A previous study demonstrated the analgesic efficacy of ketamine in patients undergoing modified pectoral nerve block in breast cancer surgery as evidenced by prolonged time to first rescue analgesia and reduced total opioid consumption.

Neostigmine has been used as an additive to local anesthetics to prolong the analgesic effect. Although there is good evidence for a spinal action of neostigmine, its analgesic efficacy as an adjuvant to local anesthetic is still unclear.

The aim of this study is to Investigate the analgesic efficacy of adding ketamine compared to neostigmine to local anesthetic in Ultrasound guided Serratus anterior plane block for patients undergoing Modified Radical Mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* ● Female patients

  * Type of surgery; Modified Radical Mastectomy (MRM).
  * Physical status ASA II, III.
  * Age ≥ 21 and ≤ 65 Years.
  * Body mass index (BMI): > 20 kg/m2 and < 35 kg/m2.

Exclusion Criteria:

* ● Patients with Known sensitivity or contraindication to drug used in the study (local anesthetics, opioids).

  * History of psychological disorders and/or chronic pain.
  * Contraindication to regional anesthesia e.g. local sepsis, pre- existing peripheral neuropathies and coagulopathy.
  * Infection of the skin at the site of needle puncture area
  * Patient refusal.
  * Severe respiratory or cardiac disorders.
  * Advanced liver or kidney disease.
  * Pregnancy.
  * Patient with surgery duration more than two hours

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-09-05 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Time of first request of analgesia | 24 hours postoperative
  it will be calculated from the time of complete injection of local anesthetics till the numerical rating scale (NRS) is ≥3.

SECONDARY OUTCOMES:
The total amount of morphine consumption | 24 hours postoperative
  Rescue analgesia will be provided in the form of IV morphine 3 mg boluses if the patient indicates Numeric Pain Rating Scale ≥ 3. The total amount of morphine given in 24 hours will be recorded for the three groups.
Total amount of intraoperative fentanyl. | 2 hours
  Rescue analgesia of fentanyl 1 μg/kg will be given if the mean arterial blood pressure or heart rate rises above 20% of baseline levels.
Numeric Pain Rating Scale | 24 hours
  A numerical rating scale (NRS) requires the patient to rate their pain on a defined scale. For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Bassant abdelhamid, M.D., Principal Investigator — Cairo University
Locations (1):
- Faculty of medicine-Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] El Mourad MB, Amer AF. Effects of adding dexamethasone or ketamine to bupivacaine for ultrasound-guided thoracic paravertebral block in patients undergoing modified radical mastectomy: A prospective randomized controlled study. Indian J Anaesth. 2018 Apr;62(4):285-291. doi: 10.4103/ija.IJA_791_17. PMID 29720754
- [Background] Pandey V, Mohindra BK, Sodhi GS. Comparative evaluation of different doses of intrathecal neostigmine as an adjuvant to bupivacaine for postoperative analgesia. Anesth Essays Res. 2016 Sep-Dec;10(3):538-545. doi: 10.4103/0259-1162.180779. PMID 27746548
- [Background] Blanco R, Parras T, McDonnell JG, Prats-Galino A. Serratus plane block: a novel ultrasound-guided thoracic wall nerve block. Anaesthesia. 2013 Nov;68(11):1107-13. doi: 10.1111/anae.12344. Epub 2013 Aug 7. PMID 23923989